CLINICAL TRIAL: NCT02945605
Title: Effects of Early Vestibular Rehabilitation Compared to Standard Care in Patients With Dizziness and Balance Disorders After Sport and Recreation Concussion
Brief Title: Effects of Early Vestibular Rehabilitation in Patients With Dizziness and Balance Disorders After Sport Concussion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of recruitment challenges
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Bara Alsalaheen, PT, Ph.D., Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00109407
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Vestibular Rehabilitation (Experimental): Participants in this group will receive a customized vestibular rehabilitation program designed and implemented by a vestibular physical therapist. The vestibular physical therapy must be initiated within 72 hours after randomization. Participants in this group will continue to receive standard of care treatment as directed by their physician.
  Interventions: Other: Early Vestibular Rehabilitation; Other: Standard of Care
- Standard of Care (Active Comparator): Participants in this group will receive standard care as directed by their physician.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Early Vestibular Rehabilitation — Two visits/week for a maximum of 5 weeks will be provided with the approximate duration for each visit estimated at 50-60 minutes. Consistent with a previously validated framework for exercise prescription in patients with concussion, the exercises provided by the treating therapist can be classified into five main exercise categories:
  1. Eye-Head coordination, gaze stability and convergence exercises
  2. Sitting balance
  3. Standing static balance (i.e. feet-in-place)
  4. Dynamic balance (feet moving, but not walking)
  5. Ambulation (gait exercises)
  6. Other exercises: Sport specific exercises, Canalith repositioning maneuvers are recorded as others
  Arms: Early Vestibular Rehabilitation
Other: Standard of Care — Standard care as directed by a physician.

SUMMARY:
This study examines the effect of early vestibular rehabilitation on reducing physical post-concussion symptoms (e.g. dizziness, balance problems) and improving the timeline to achieve medical clearance to return to activities such as sports and work activities. Half of the participants will receive early vestibular rehabilitation added to standard of care, while the other half will receive standard of care only.

DETAILED DESCRIPTION:
As awareness of concussion and the numbers of reported concussions increase every year in the last few years, so does the need for more effective treatment strategies. Concussions can lead to a variety of symptoms that may last from days to weeks after injury.[1] Dizziness and vestibular impairments are prevalent in up to 81% of patients after concussion.[2,3] Additionally, dizziness and vestibular impairments are predictive of prolonged recovery times after concussion.[4] Although there are few studies suggesting that vestibular rehabilitation after concussion is promising,[5,6] there continues to be a void in well-controlled studies verifying that vestibular rehabilitation can be used to treat patients with dizziness and balance disorders after concussion. Due to the lack of controlled studies and current practice patterns, patients with concussions are not seen for physical therapy until weeks or months after their injury. The purpose of this study is to examine the effect of early vestibular rehabilitation on reducing physical post-concussion symptoms (e.g. dizziness, balance problems), and improving the timeline to achieve medical clearance to return to activities such as sports and work activities, when compared to STANDARD care. The findings of this study are expected to provide medical and sports related professionals with appropriate concussion treatment strategies and improve outcomes of patients suffering from concussion.

ELIGIBILITY:
Inclusion Criteria:

* Dizziness or balance problems within 10 days of concussion

Exclusion Criteria:

* None

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Change in Sports Concussion Assessment Tool (SCATIII) Symptom Inventory | At every 7 days since concussion and the end of the study (up to 5 weeks, or after full resolution of symptoms, whichever occurs first)
  The change is calculated by subtracting the score obtained at a designated time point from the initial score.

SECONDARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) | At every 7 days since concussion and the end of the study (up to 5 weeks, or after full resolution of symptoms, whichever occurs first)
  The DHI assesses the individual's handicap due to their dizziness problem in 25 items relating to physical, emotional, and functional domains. The highest overall score of the test is 100 with higher scores indicating greater dizziness handicap. Participants who are 18 years or older on the initial assessment day will complete the original DHI, and participants younger than 18 will complete the adolescents version of DHI.
  The change is calculated by subtracting the score obtained at a designated time point from the initial score.
Global Rating of Change (GRC) | At every 7 days since concussion and the end of the study (up to 5 weeks, or after full resolution of symptoms, whichever occurs first)
  GRC scales ask that a person assess his or her current health status, recall that status at a previous time-point, and then calculate the difference between the two. The scoring ranges from "A very great deal worse (-7)" to "A very great deal better (7)."
Change in Vestibular Ocular Motor Screening (VOMS) | Up to 5 weeks, or after full resolution of symptoms, whichever occurs first
  Participants will complete the VOMS testing seven items: smooth pursuit, saccades (horizontal and vertical), vestibulo-ocular reflex (VOR) (horizontal and vertical), vision motion sensitivity testing, and Near-Point-of-Convergence (NPC) distance (three trials). Participants are asked to report the intensity, using a scale from 0 (none) -10 (severe), of four possible symptoms (headache, dizziness, nausea, and fogginess). The participant reports at baseline and after each of the seven VOMS tests. Any change in each of the four symptoms from baseline is reported for each of the seven VOMS items. The total symptom score is calculated by summating any change in four symptoms from baseline for each of the seven VOMS tests.
  The change is calculated by subtracting the score obtained at the termination of the study from the initial score.
Change in Functional Gait Assessment (FGA) | Up to 5 weeks, or after full resolution of symptoms, whichever occurs first
  The FGA assesses the ability to walk with head turns, changes of speed, pivot turns, backwards and narrow base of support. The scale for each item ranges from 0-3, where 0 means severe impairment and 3 means normal. The highest possible score is 30. Higher scores indicate better performance.
  The change is calculated by subtracting the score obtained at the termination of the study from the initial score.
Change in Original and Cognitive Timed Up & Go (TUG) | Up to 5 weeks, or after full resolution of symptoms, whichever occurs first
  The TUG is a timed test during which the participant stands from a chair, walks three meters at their normal walking speed, returns to the chair, and sits down. The cognitive TUG is completed while counting backwards in threes from a random start point. An automaticity index is calculated to assess the impact of both dual tasks. The speed under the dual-task condition is expressed as a percentage of the speed under the single-task condition: (single task/dual task) *100. A maximal achievable score of 100% indicated no decrease in performance under the dual-task condition. This index is developed as a method for standardizing the assessment of dual-task performance and its effect on automaticity.
  The change is calculated by subtracting the score obtained at the termination of the study from the initial score.
Change in Clinical Dynamic Visual Acuity | Up to 5 weeks, or after full resolution of symptoms, whichever occurs first
  First perform the test for static visual acuity: patient may wear glasses or contacts. Have patient sit/stand about 10 feet away from eye chart (LogMAR). Have them read the lowest line they can see until they cannot correctly identify all the letters in a given line. Note which line this is. Dynamic Visual Acuity: Stand behind patient and tilt their head down 20°. Rotate their head at 2 Hz (240 beats/min on metronome) and have them read the lowest line possible until they cannot correctly identify all the letters in a given line. Note which line this is. Abnormal Test: greater than 2 line difference or if patient experiences dizziness which they rate on a 0 to 10 scale.
  The change is calculated by subtracting the score obtained at the termination of the study from the initial score.
Change in Original and dual task Balance Error Scoring System (BESS) | Up to 5 weeks, or after full resolution of symptoms, whichever occurs first
  Participants will perform the BESS while on a NeuroCom® portable force plate system. Participants are asked to stand on the force plate and maintain balance with eyes closed and hands on their iliac crests under 6 different conditions (20 seconds each):
  1. firm surface, feet together
  2. firm surface, single leg stance
  3. firm surface, tandem stance
  4. foam surface, feet together
  5. foam surface, single leg stance
  6. foam surface, tandem stance
  This procedure allows for simultaneous computation of sway by the force plate and clinical assessment of balance errors as indicated by the BESS.
  For the dual task Balance Error Scoring System, the BESS will be completed as per BESS protocol with a cognitive task of serial threes. For the serial threes task, participants are given a random number between 80 and 100 and instructed to subtract by threes. When participants fail to perform a correct subtraction, it is considered an error.
Change in Limits of Stability (LOS) Test | Up to 5 weeks, or after full resolution of symptoms, whichever occurs first
  The LOS quantifies the maximum distance the patient can intentionally displace their Center of Gravity (COG) in the four cardinal directions and the four diagonal directions, and maintain stability at those positions. Measured parameters are reaction time, COG movement velocity, directional control, end point excursion, and maximum excursion.
  The change is calculated by subtracting the score obtained at the termination of the study from the initial score.
Time until medical clearance to return to sports/activities | The number of days between concussion and the day when a physician provided full clearance to return to sport/activities (retrieved from medical record) up to 52 weeks from concussion date. [the date of clearance - the concussion date]
  The number of days between concussion and the day when a physician provided full clearance to return to sport/activities

CONTACTS AND LOCATIONS:
Overall Officials: Bara Alsalaheen, PT, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broglio SP, Cantu RC, Gioia GA, Guskiewicz KM, Kutcher J, Palm M, Valovich McLeod TC; National Athletic Trainer's Association. National Athletic Trainers' Association position statement: management of sport concussion. J Athl Train. 2014 Mar-Apr;49(2):245-65. doi: 10.4085/1062-6050-49.1.07. Epub 2014 Mar 7. PMID 24601910
- [Background] Zhou G, Brodsky JR. Objective vestibular testing of children with dizziness and balance complaints following sports-related concussions. Otolaryngol Head Neck Surg. 2015 Jun;152(6):1133-9. doi: 10.1177/0194599815576720. Epub 2015 Mar 27. PMID 25820582
- [Background] Corwin DJ, Wiebe DJ, Zonfrillo MR, Grady MF, Robinson RL, Goodman AM, Master CL. Vestibular Deficits following Youth Concussion. J Pediatr. 2015 May;166(5):1221-5. doi: 10.1016/j.jpeds.2015.01.039. Epub 2015 Mar 5. PMID 25748568
- [Background] Lau BC, Kontos AP, Collins MW, Mucha A, Lovell MR. Which on-field signs/symptoms predict protracted recovery from sport-related concussion among high school football players? Am J Sports Med. 2011 Nov;39(11):2311-8. doi: 10.1177/0363546511410655. Epub 2011 Jun 28. PMID 21712482
- [Background] Alsalaheen BA, Mucha A, Morris LO, Whitney SL, Furman JM, Camiolo-Reddy CE, Collins MW, Lovell MR, Sparto PJ. Vestibular rehabilitation for dizziness and balance disorders after concussion. J Neurol Phys Ther. 2010 Jun;34(2):87-93. doi: 10.1097/NPT.0b013e3181dde568. PMID 20588094
- [Background] Schneider KJ, Meeuwisse WH, Nettel-Aguirre A, Barlow K, Boyd L, Kang J, Emery CA. Cervicovestibular rehabilitation in sport-related concussion: a randomised controlled trial. Br J Sports Med. 2014 Sep;48(17):1294-8. doi: 10.1136/bjsports-2013-093267. Epub 2014 May 22. PMID 24855132